CLINICAL TRIAL: NCT04567459
Title: The Effect of Nutrition for the Colorectal Cancer Patients Receiving Chemotherapy-randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Hanben Enterprise (Unknown)
Responsible Party: Principal Investigator, Wan-Hsiang Hu, Attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202000035A3
Record Dates: First submitted 2020-08-26; First posted 2020-09-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Chemotherapy; Nutrition; Sarcopenia
MeSH Terms: conditions — Colorectal Neoplasms; Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group: chemotherapy (No Intervention): No intervention
- experimental group: chemotherapy and nutrition support (Experimental): Premium amino acids 1pc bid for 6 months
  Interventions: Dietary Supplement: Premium Amino Acids

INTERVENTIONS:
Dietary Supplement: Premium Amino Acids — after Chemotherapy ang surgery one pack of Premium Amino Acids in the morning and evening
  Arms: experimental group: chemotherapy and nutrition support

SUMMARY:
We use clinical trial to explore the effect of nutrition support in colorectal cancer patients receiving postoperative adjuvant chemotherapy.

DETAILED DESCRIPTION:
Colorectal cancer is the most common cancer in Taiwan. Side effects induced by postoperative adjuvant chemotherapy will affect nutrition status and may delay treatment and affect prognosis. Sarcopenia may be noted in some patients and increase the toxicities of chemotherapy. The studies of intervention include nutrition consultant and treatment like protein, fish oil or Vitamin D supplement. Premium amino acids include multiple amino acids and organic Selenium and have effect in inhibition of tumor proliferation according to colorectal cancer cell and animal experiments.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20
* Radical operation for stage III and stage II with high risk colorectal cancer
* Agree to join the trial and sign the informed consent form

Exclusion Criteria:

* Unable to receive chemotherapy
* Unstable vital sign
* Not suitable after evaluation by Principal Investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-27 (Estimated); Primary Completion 2021-02-22 (Estimated); Study Completion 2021-02-22 (Estimated)

PRIMARY OUTCOMES:
Assessment of adverse event | 2 weeks after chemotherapy
  Evaluation of adverse event(Grade 1-4) between control group and experimental group before every chemotherapy(total 12 times)
1)Nutrition assessment | 2 weeks after chemotherapy
  albumin level between two group before every chemotherapy(total 12 times)
2)Nutrition assessment | 2 weeks after chemotherapy
  pre-albumin level between two group before every chemotherapy(total 12 times)
1)Sarcopenia assessment muscle power | At 1st cycle of chemotherapy (each cycle is 2 weeks).
  1-1)Assessment with Grip strength(Kg)
1)Sarcopenia assessment muscle power | At 12th cycle of chemotherapy (each cycle is 2 weeks).
  1-2)Assessment with Grip strength(Kg)
2)Sarcopenia assessment muscle power | At 1st cycle of chemotherapy (each cycle is 2 weeks).
  2-1)Assessment with ASM/heigh2(Kg/m2)
2)Sarcopenia assessment muscle power | At 12st cycle of chemotherapy (each cycle is 2 weeks).
  2-2)Assessment with ASM/heigh2(Kg/m2)
3)Sarcopenia assessment | At 1st cycle of chemotherapy (each cycle is 2 weeks).
  3-1)Assessment with speed(m/s)
3)Sarcopenia assessment | At 12th cycle of chemotherapy (each cycle is 2 weeks).
  3-2)Assessment with speed(m/s)
4)Sarcopenia assessment | At 1st cycle of chemotherapy (each cycle is 2 weeks).
  4-1)Assessment with DXA(g/cm2)
4)Sarcopenia assessment | At 12th cycle of chemotherapy (each cycle is 2 weeks).
  4-2)Assessment with DXA(g/cm2)
5)Sarcopenia assessment | At 6th cycle of chemotherapy (each cycle is 2 weeks).
  5-1)Assessment with abdominal CT
5)Sarcopenia assessment | At 12th cycle of chemotherapy (each cycle is 2 weeks).
  5-2)Assessment with abdominal CT

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital,Kaohsiung, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Chiang CJ, Lo WC, Yang YW, You SL, Chen CJ, Lai MS. Incidence and survival of adult cancer patients in Taiwan, 2002-2012. J Formos Med Assoc. 2016 Dec;115(12):1076-1088. doi: 10.1016/j.jfma.2015.10.011. Epub 2016 Jan 16. PMID 26786251
- [Background] Andre T, Boni C, Navarro M, Tabernero J, Hickish T, Topham C, Bonetti A, Clingan P, Bridgewater J, Rivera F, de Gramont A. Improved overall survival with oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment in stage II or III colon cancer in the MOSAIC trial. J Clin Oncol. 2009 Jul 1;27(19):3109-16. doi: 10.1200/JCO.2008.20.6771. Epub 2009 May 18. PMID 19451431
- [Background] Casadaban L, Rauscher G, Aklilu M, Villenes D, Freels S, Maker AV. Adjuvant chemotherapy is associated with improved survival in patients with stage II colon cancer. Cancer. 2016 Nov 15;122(21):3277-3287. doi: 10.1002/cncr.30181. Epub 2016 Jul 15. PMID 27417445
- [Background] Gelibter AJ, Caponnetto S, Urbano F, Emiliani A, Scagnoli S, Sirgiovanni G, Napoli VM, Cortesi E. Adjuvant chemotherapy in resected colon cancer: When, how and how long? Surg Oncol. 2019 Sep;30:100-107. doi: 10.1016/j.suronc.2019.06.003. Epub 2019 Jul 2. PMID 31500770
- [Background] Jung HW, Kim JW, Kim JY, Kim SW, Yang HK, Lee JW, Lee KW, Kim DW, Kang SB, Kim KI, Kim CH, Kim JH. Effect of muscle mass on toxicity and survival in patients with colon cancer undergoing adjuvant chemotherapy. Support Care Cancer. 2015 Mar;23(3):687-94. doi: 10.1007/s00520-014-2418-6. Epub 2014 Aug 28. PMID 25163434
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Bano G, Trevisan C, Carraro S, Solmi M, Luchini C, Stubbs B, Manzato E, Sergi G, Veronese N. Inflammation and sarcopenia: A systematic review and meta-analysis. Maturitas. 2017 Feb;96:10-15. doi: 10.1016/j.maturitas.2016.11.006. Epub 2016 Nov 13. PMID 28041587
- [Background] Lin JX, Lin JP, Xie JW, Wang JB, Lu J, Chen QY, Cao LL, Lin M, Tu R, Zheng CH, Huang CM, Li P. Prognostic Value and Association of Sarcopenia and Systemic Inflammation for Patients with Gastric Cancer Following Radical Gastrectomy. Oncologist. 2019 Nov;24(11):e1091-e1101. doi: 10.1634/theoncologist.2018-0651. Epub 2019 Mar 25. PMID 30910865
- [Background] Tessier AJ, Chevalier S. An Update on Protein, Leucine, Omega-3 Fatty Acids, and Vitamin D in the Prevention and Treatment of Sarcopenia and Functional Decline. Nutrients. 2018 Aug 16;10(8):1099. doi: 10.3390/nu10081099. PMID 30115829
- [Background] Mazzuca F, Roberto M, Arrivi G, Sarfati E, Schipilliti FM, Crimini E, Botticelli A, Di Girolamo M, Muscaritoli M, Marchetti P. Clinical Impact of Highly Purified, Whey Proteins in Patients Affected With Colorectal Cancer Undergoing Chemotherapy: Preliminary Results of a Placebo-Controlled Study. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419866920. doi: 10.1177/1534735419866920. PMID 31370717